CLINICAL TRIAL: NCT04061343
Title: The Effects of chaNging LIGHT Levels on Contrast sENsitivity in Patients With Glaucoma
Acronym: ENLIGHTEN
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2017/95
Record Dates: First submitted 2019-05-03; First posted 2019-08-19 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective observational study where participants will be recruited from the Ophthalmology department (Outpatient department, Eye Casualty). Only one research visit will be required. Participants will be asked to fill in a set of questionnaires (Visual Functioning Questionnaire-15(61), Low Luminance Questionnaire(62)) assessing their quality of life and vision and their full medical history will be collected. Then they will have their contrast sensitivity tested under various light conditions. If a recent visual field test is not available, that might be performed as part of the study.

DETAILED DESCRIPTION:
The purpose of our, real world study is to explore contrast sensitivity differences after changes in ambient light setting in patients with glaucoma compared with controls (patients with ocular hypertension). Participants will be asked to read a Pelli- Robson chart under photopic (bright light conditions) and mesopic (intermediate light conditions); followed by scotopic conditions (dim light conditions). This chart is a fast, easy, and effective way to measure spatial contrast sensitivity with reliable and reproducible results(60). This study will therefore help clinicians gain more insight into glaucoma related disability and provide a possible additional tool to visual field testing in patients with advanced glaucoma where VF testing may be hampered by floor effects.

ELIGIBILITY:
Inclusion Criteria:

* • Male or Female, aged 40 years or above.

  * Diagnosis of glaucoma (including primary open angle glaucoma, pigment dispersion syndrome, pseudoexfoliation, normal tension glaucoma, chronic angle closure glaucoma, narrow angle glaucoma) or ocular hypertension
  * Willing and able to give informed consent for participation in the study.
  * Best Corrected Visual Acuity equal or better than 6/12 as measured with the Snellen Chart

Exclusion Criteria:

* • Neovascular, uveitic, acute angle closure glaucoma

  * Non-glaucomatous ocular disease such as AMD, Diabetic retinopathy, Inherited eye diseases
  * Visually significant cataracts (Distance VA ≤ 6/12 (0.30 LogMAR) and grade ≥ grade 2 nuclear sclerosis.)
  * Current use of miotic glaucoma medication
  * Incisional or laser eye surgery within 3 months of enrolment
  * Severely impaired cognition
  * Self-reported physical ability limiting function (e.g. stroke)
  * Unreliable visual fields (SITA Standard or SITA Fast: fixation losses >20% or false-positive errors >33% or false-negative errors >33%)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of glaucoma (including primary open angle glaucoma, pigment dispersion syndrome, pseudoexfoliation, normal tension glaucoma, chronic angle closure glaucoma, narrow angle glaucoma) or ocular hypertension aged ≥40 years old.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
vision-related quality of life in patients with glaucoma | 1 day study visit
  assessed using the the visual functioning questionnaire - 25 questionnaire
Visual function | through study completion, an average of 1 year
  assessed using the low luminance questionnaire

SECONDARY OUTCOMES:
To correlate visual impairment with contrast sensitivity results | through study completion, an average of 1 year
  measured with Quality of Life questionnaires (Visual Functioning Questionnaire-25, Low Luminance Questionnaire)
Contrast Sensitivitiy | through study completion, an average of 1 year
  Participants' contrast sensitivity will be tested under photopic (bright light conditions), mesopic (intermediate light conditions) and/or scotopic conditions (dim light conditions).

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom